CLINICAL TRIAL: NCT02060162
Title: Antiretroviral Treatment Outcomes in HIV-HBV Co-infected Patients in Southern Africa: a Collaborative Multi-country Prospective Cohort Analysis for International Epidemiologic Databases to Evaluate AIDS- Southern Africa (HIV/HBV-coinfection in IeDEA-SA)
Brief Title: Antiretroviral Treatment Outcomes in HIV-HBV Co-infected Patients in Southern Africa
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Michael Vinikoor, Associate Professor, University of Alabama at Birmingham
Other Study IDs: F160229001
Record Dates: First submitted 2014-02-09; First posted 2014-02-11 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis B Virus; HIV; Antiretroviral Therapy; Africa; Liver Fibrosis; Alcohol Use Disorder
Keywords: antiretroviral therapy; Hepatitis C virus
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; Alcoholism; Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimen storage is optional and participants will provide additional informed consent. The laboratory will store leftover blood specimens for up to 5 years for hepatitis related serologic, immunological, and virologic studies pending availability of funding. Use of specimens for any tests outside the realm of the goals and objectives of this study will require additional approval by the Zambian IRB.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV/HBV co-infected: 150-200 patients in Zambia and 250-300 across all sites
  Interventions: Other: Standard of care
- HIV mono-infected: 700-750 patients in Zambia and 1600-1700 across all sites
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — routine standard of care per Ministry of Health protocol including blood draws and examinations.

SUMMARY:
This is a prospective HIV cohort that aims to establish causes of liver disease among HIV-infected individuals in Zambia, including viral hepatitis and alcohol.

DETAILED DESCRIPTION:
The study will take place during routinely scheduled ART visits as per Ministry of Health guidelines. Routinely collected programmatic data will be used to assess general HIV outcomes (CD4 response, loss to follow-up, death) as well as collecting study specific data (hepatitis testing, questionnaire regarding risk factors for hepatitis/liver disease, and non-invasive liver scan) to address other aims. The study will be implemented at two sites in Southern Africa (Zambia and Mozambique) with a total enrollment across all sites of 1,900 participants. The Zambia site will only enroll 900.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Male or female aged ≥18 years
* ART naïve
* ART eligible as defined by Zambian or WHO treatment guidelines
* Initiating an ART regimen including at least 3 drugs at one of the study sites.
* Willing to provide signed informed consent and be followed at the clinical site.

Exclusion Criteria:

* Patients who are not planning to remain in the catchment area from which they were recruited for the duration of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of 1,900 consecutive patients starting ART (900 in Zambia and 1,000 in Mozambique) is planned.
Sampling Method: Non-Probability Sample
Enrollment: 897 (Actual)
Dates: Start 2013-10; Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Immunological response | 12 months post enrollment
  A linear mixed effect model will be used to evaluate immunological response to ART in patients with and without viral hepatitis

SECONDARY OUTCOMES:
HIV virological response | 12 months post enrollment
  Virological response will be evaluated using Cox regression analyses.
Mortality | 12 months
  Deaths will be ascertained
Hepatotoxicity events | 6 and 12 months
  These events will be defined as an increase in the level of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 time the upper limit within the first year of ART.
Prevalence liver fibrosis | Baseline and one year after start of ART
  The prevalence of liver fibrosis will be measured to compare HIV/hepatitis coinfected versus HIV monoinfected patients using transient elastography.
HBV drug resistance | 1 and 2 years post enrollment
  The presence of HBV drug resistance in co-infected patients who fail treatment after 1 year will be measured
Incidence of HBV infection | 12 and 24 months post enrollment
  The incidence of HBV infection during ART will be measured.
Prevalence of HIV/HCV coinfection | Baseline
  Describe prevalence of coinfection at ART initiation
Alcohol use patterns | Baseline, 12, and 24 months
  Describe the proportion with unhealthy levels of drinking before and after ART

CONTACTS AND LOCATIONS:
Overall Officials: Roma Chilengi, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia; Michael Vinikoor, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Barth RE, Huijgen Q, Taljaard J, Hoepelman AI. Hepatitis B/C and HIV in sub-Saharan Africa: an association between highly prevalent infectious diseases. A systematic review and meta-analysis. Int J Infect Dis. 2010 Dec;14(12):e1024-31. doi: 10.1016/j.ijid.2010.06.013. Epub 2010 Sep 25. PMID 20870439
- [Background] Chang TT, Gish RG, de Man R, Gadano A, Sollano J, Chao YC, Lok AS, Han KH, Goodman Z, Zhu J, Cross A, DeHertogh D, Wilber R, Colonno R, Apelian D; BEHoLD AI463022 Study Group. A comparison of entecavir and lamivudine for HBeAg-positive chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1001-10. doi: 10.1056/NEJMoa051285. PMID 16525137
- [Background] Davies J, van Oosterhout JJ, Nyirenda M, Bowden J, Moore E, Hart IJ, Zijlstra EE, Chaponda M, Faragher B, Beeching NJ, Beadsworth MB. Reliability of rapid testing for hepatitis B in a region of high HIV endemicity. Trans R Soc Trop Med Hyg. 2010 Feb;104(2):162-4. doi: 10.1016/j.trstmh.2009.10.010. PMID 19931107
- [Background] De Luca A, Bugarini R, Lepri AC, Puoti M, Girardi E, Antinori A, Poggio A, Pagano G, Tositti G, Cadeo G, Macor A, Toti M, D'Arminio Monforte A; Italian Cohort Naive Antiretrovirals Study Group. Coinfection with hepatitis viruses and outcome of initial antiretroviral regimens in previously naive HIV-infected subjects. Arch Intern Med. 2002 Oct 14;162(18):2125-32. doi: 10.1001/archinte.162.18.2125. PMID 12374521
- [Background] Di Bisceglie AM, Maskew M, Schulze D, Reyneke A, McNamara L, Firnhaber C. HIV-HBV coinfection among South African patients receiving antiretroviral therapy. Antivir Ther. 2010;15(3 Pt B):499-503. doi: 10.3851/IMP1494. PMID 20516571
- [Background] Dienstag JL, Schiff ER, Wright TL, Perrillo RP, Hann HW, Goodman Z, Crowther L, Condreay LD, Woessner M, Rubin M, Brown NA. Lamivudine as initial treatment for chronic hepatitis B in the United States. N Engl J Med. 1999 Oct 21;341(17):1256-63. doi: 10.1056/NEJM199910213411702. PMID 10528035
- [Background] Firnhaber C, Reyneke A, Schulze D, Malope B, Maskew M, MacPhail P, Sanne I, Di Bisceglie A. The prevalence of hepatitis B co-infection in a South African urban government HIV clinic. S Afr Med J. 2008 Jul;98(7):541-4. PMID 18785395
- [Background] Hoffmann CJ, Charalambous S, Martin DJ, Innes C, Churchyard GJ, Chaisson RE, Grant AD, Fielding KL, Thio CL. Hepatitis B virus infection and response to antiretroviral therapy (ART) in a South African ART program. Clin Infect Dis. 2008 Dec 1;47(11):1479-85. doi: 10.1086/593104. PMID 18937580
- [Background] Hoffmann CJ, Charalambous S, Thio CL, Martin DJ, Pemba L, Fielding KL, Churchyard GJ, Chaisson RE, Grant AD. Hepatotoxicity in an African antiretroviral therapy cohort: the effect of tuberculosis and hepatitis B. AIDS. 2007 Jun 19;21(10):1301-8. doi: 10.1097/QAD.0b013e32814e6b08. PMID 17545706
- [Background] KASOLO, F. (2003) Hepatitis B virus infection in human immunodeficiency virus seropositive patients at the University Teaching Hospital, Lusaka, Zambia: Interrelationship. IN SAKALA, I. (Ed.) Abstract no. B12601. The XV International Aids Conference, International Aids Society.
- [Background] Kwon H, Lok AS. Hepatitis B therapy. Nat Rev Gastroenterol Hepatol. 2011 May;8(5):275-84. doi: 10.1038/nrgastro.2011.33. Epub 2011 Mar 22. PMID 21423260
- [Background] Lok AS, Lai CL, Leung N, Yao GB, Cui ZY, Schiff ER, Dienstag JL, Heathcote EJ, Little NR, Griffiths DA, Gardner SD, Castiglia M. Long-term safety of lamivudine treatment in patients with chronic hepatitis B. Gastroenterology. 2003 Dec;125(6):1714-22. doi: 10.1053/j.gastro.2003.09.033. PMID 14724824
- [Background] Lok AS, Zoulim F, Locarnini S, Bartholomeusz A, Ghany MG, Pawlotsky JM, Liaw YF, Mizokami M, Kuiken C; Hepatitis B Virus Drug Resistance Working Group. Antiviral drug-resistant HBV: standardization of nomenclature and assays and recommendations for management. Hepatology. 2007 Jul;46(1):254-65. doi: 10.1002/hep.21698. PMID 17596850
- [Background] Marcellin P, Heathcote EJ, Buti M, Gane E, de Man RA, Krastev Z, Germanidis G, Lee SS, Flisiak R, Kaita K, Manns M, Kotzev I, Tchernev K, Buggisch P, Weilert F, Kurdas OO, Shiffman ML, Trinh H, Washington MK, Sorbel J, Anderson J, Snow-Lampart A, Mondou E, Quinn J, Rousseau F. Tenofovir disoproxil fumarate versus adefovir dipivoxil for chronic hepatitis B. N Engl J Med. 2008 Dec 4;359(23):2442-55. doi: 10.1056/NEJMoa0802878. PMID 19052126
- [Background] Nagu TJ, Bakari M, Matee M. Hepatitis A, B and C viral co-infections among HIV-infected adults presenting for care and treatment at Muhimbili National Hospital in Dar es Salaam, Tanzania. BMC Public Health. 2008 Dec 19;8:416. doi: 10.1186/1471-2458-8-416. PMID 19099553
- [Background] Nikolopoulos GK, Paraskevis D, Hatzitheodorou E, Moschidis Z, Sypsa V, Zavitsanos X, Kalapothaki V, Hatzakis A. Impact of hepatitis B virus infection on the progression of AIDS and mortality in HIV-infected individuals: a cohort study and meta-analysis. Clin Infect Dis. 2009 Jun 15;48(12):1763-71. doi: 10.1086/599110. PMID 19435436
- [Background] Nyirenda M, Beadsworth MB, Stephany P, Hart CA, Hart IJ, Munthali C, Beeching NJ, Zijlstra EE. Prevalence of infection with hepatitis B and C virus and coinfection with HIV in medical inpatients in Malawi. J Infect. 2008 Jul;57(1):72-7. doi: 10.1016/j.jinf.2008.05.004. Epub 2008 Jun 13. PMID 18555534
- [Background] Oshitani H, Kasolo F, Tembo C, Mpabalwani M, Mizuta K, Luo N, Suzuki H, Numazaki Y. Hepatitis B virus infection among pregnant women in Zambia. East Afr Med J. 1995 Dec;72(12):813-5. PMID 8689985
- [Background] Otegbayo JA, Taiwo BO, Akingbola TS, Odaibo GN, Adedapo KS, Penugonda S, Adewole IF, Olaleye DO, Murphy R, Kanki P. Prevalence of hepatitis B and C seropositivity in a Nigerian cohort of HIV-infected patients. Ann Hepatol. 2008 Apr-Jun;7(2):152-6. PMID 18626434
- [Background] Stabinski L, Reynolds SJ, Ocama P, Laeyendecker O, Ndyanabo A, Kiggundu V, Boaz I, Gray RH, Wawer M, Thio C, Thomas DL, Quinn TC, Kirk GD; Rakai Health Sciences Program. High prevalence of liver fibrosis associated with HIV infection: a study in rural Rakai, Uganda. Antivir Ther. 2011;16(3):405-11. doi: 10.3851/IMP1783. PMID 21555823
- [Background] Selabe SG, Lukhwareni A, Song E, Leeuw YG, Burnett RJ, Mphahlele MJ. Mutations associated with lamivudine-resistance in therapy-naive hepatitis B virus (HBV) infected patients with and without HIV co-infection: implications for antiretroviral therapy in HBV and HIV co-infected South African patients. J Med Virol. 2007 Nov;79(11):1650-4. doi: 10.1002/jmv.20974. PMID 17854040
- [Background] Wiersma ST, McMahon B, Pawlotsky JM, Thio CL, Thursz M, Lim SG, Ocama P, Esmat G, Mendy M, Bell D, Vitoria M, Eramova I, Lavanchy D, Dusheiko G; World Health Organization Department of Immunization, Vaccines and Biologicals. Treatment of chronic hepatitis B virus infection in resource-constrained settings: expert panel consensus. Liver Int. 2011 Jul;31(6):755-61. doi: 10.1111/j.1478-3231.2010.02373.x. Epub 2011 Feb 15. PMID 21645206
- [Derived] Vinikoor MJ, Sinkala E, Chilengi R, Mulenga LB, Chi BH, Zyambo Z, Hoffmann CJ, Saag MS, Davies MA, Egger M, Wandeler G; IeDEA- Southern Africa. Impact of Antiretroviral Therapy on Liver Fibrosis Among Human Immunodeficiency Virus-Infected Adults With and Without HBV Coinfection in Zambia. Clin Infect Dis. 2017 May 15;64(10):1343-1349. doi: 10.1093/cid/cix122. PMID 28158504
- See also: University of North Carolina website — http://www.unc.edu